CLINICAL TRIAL: NCT05352425
Title: A Study Assessing the Effect of the MobiusHD® Implant in Renal Hemodialysis Subjects Presented With Uncontrolled Hypertension
Brief Title: Effect of the MobiusHD® in Renal Hemodialysis Subjects With Uncontrolled Hypertension
Acronym: HD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decided to not pursue study at this time
Sponsor: Vascular Dynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRD0597, CRD0597_CAN
Record Dates: First submitted 2022-04-01; First posted 2022-04-28 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Uncontrolled Hypertension
Keywords: Uncontrolled Hypertension; End Stage Renal Disease; MobiusHD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- MobiusHD (Experimental): Each subject enrolled in the study will undergo implantation of the MobiusHD® device
  Interventions: Device: MobiusHD

INTERVENTIONS:
Device: MobiusHD — The MobiusHD® device is a nickel-titanium device that is implanted in the internal carotid sinus using a minimally invasive approach.

SUMMARY:
This is a prospective, multi-center, open-label clinical trial intended to evaluate the safety and benefit of the MobiusHD® system in renal hemodialysis subjects with uncontrolled hypertension.

DETAILED DESCRIPTION:
Renal hemodialysis patients with uncontrolled hypertension will be considered for the study. Subjects who meet initial screening requirements will undergo non-invasive imaging of the carotid anatomy to assess adequacy of the anatomy to allow placement of the MobiusHD® device. Eligible subjects will receive an implant placed in the internal carotid artery.

Following implantation of the device, subjects will be followed for 60 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 years or above
2. End Stage Renal Disease subjects receiving renal hemodialysis at least 3 months prior to procedure
3. Hypertension that is unresponsive to medical therapy of at least 3 anti-hypertensive medication classes
4. Deemed an acceptable candidate for the implant procedure by the investigator
5. Adequacy of the carotid anatomy for treatment with the MobiusHD implant based on non-invasive carotid duplex and CTA imaging, and invasive carotid angiography

Exclusion Criteria:

1. Known or clinically suspected baroreflex failure or autonomic neuropathy
2. History of intradialytic hypotension within the past 3 months
3. Secondary cause of hypertension except treated obstructive sleep apnea syndrome
4. BMI ≥ 45 kg/m2
5. Presence of atherosclerotic plaque in the intended side for implantation as determined by carotid duplex

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Incidence of intradialytic hypotension (IDH) | 6 months
  Incidence of intradialytic hypotension between baseline and 6 months
Major adverse neurological and cardiovascular events (MANCE) | 6 months
  Incidence of MANCE events between baseline and 6 months
Change in 44-hour ambulatory blood pressure measurements (ABPM) | 6 months
  Change in 44-hour ABPM between baseline and 6 months
Change in rate of blood pressure related hospitalizations | 6 months
  Change in rate of blood pressure related hospitalizations between baseline and 6 months
Change in Quality of Life (QoL), assessed by the London Evaluation of Illness (LEVIL) questionnaire | 6 months
  Changes in the London Evaluation of Illness (LEVIL) questionnaire between baseline and 6 months. The scores on the LEVIL range from 0 to 100 Units on a Scale. A higher unit score indicates a better outcome.
Change in Quality of Life (QoL), assessed by the Kidney Disease Quality of Life (KDQOL-36) questionnaire | 6 months
  Changes in the Kidney Disease Quality of Life (KDQOL-36) questionnaire between baseline and 6 months. The KDQOL-36 compares patients to others of the same age, gender, and diabetes status and is measured on by Units on a Scale. The higher a patient's average is above the mean indicates a better outcome.